CLINICAL TRIAL: NCT04091347
Title: Pilot Study of Depression and Pain Perseverance Through Empowered Recovery (DAPPER) Intervention
Brief Title: Depression and Pain Perseverance Through Empowered Recovery Intervention
Acronym: DAPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00226182; 75206 (Other Grant/Funding Number: Robert Wood Johnson Harold Amos Medical Faculty Program); P30AG021334 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pain; Depressive Symptoms; Frailty; Aging
Keywords: African American; Women's Health
MeSH Terms: conditions — Pain; Depression; Frailty

STUDY DESIGN:
Intervention Model Description: The investigator will conduct subsequent single blind wait list control design to test the preliminary effects of DAPPER and the feasibility of older African American women integrating strategies to address pain, depression, and frailty that are tailored to the individual into the individual's daily routines.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician will be responsible for randomization and the investigator and study team will not have knowledge if participants are assigned to intervention group or wait list control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention group will receive the intervention for 12 weeks. The wait list control group will have outcomes measured but will not receive the intervention at this time.
  Interventions: Behavioral: DAPPER
- Wait List Control Arm (Active Comparator): Once the intervention group has completed the intervention the wait list control group will complete the intervention.
  Interventions: Behavioral: DAPPER

INTERVENTIONS:
Behavioral: DAPPER — The DAPPER program is person directed and will consist of 8 nurse visits during which the nurse assesses each participant for pain, depression and frailty and then implements a manualized individually tailored intervention. Participants will be randomized into either the intervention or the wait list control group. Once the intervention group has completed the intervention group's visits, the wait list control group will begin the waitlist control group's visits. All participants will all be offered the same information and format of nurse visits. The nurses will systematically tailor the content of the visits to the participants' risk profile and goals based on protocols. All participants will be assessed at the start of the study, at 12 weeks and 24 weeks.

SUMMARY:
African American women who are 50 years of age and older with depressive symptoms, pain and difficulty with mobility will participate in the DAPPER intervention study that includes 8 nurse visits in participants' homes to help participants with participants' pain and mood.

DETAILED DESCRIPTION:
The proposed intervention is called Depression and Pain Perseverance through Empowered Recovery (DAPPER). The investigators are adapting the Get Busy Get Better intervention by adding components (e.g. nurse visits and person directed goals) from the CAPABLE study for this intervention. The investigator will further develop the intervention through this two-phase pilot test. The aims of this pilot project are to 1) test the Depression and Pain Perseverance through Empowered Recovery (DAPPER) program for feasibility and acceptability. Specifically, the investigators will test the effect size of DAPPER on pain and depressive symptoms from baseline to 12 weeks (compare intervention to wait list control group) and then at 24 weeks to compare the intervention group to wait list control group once again. 2) estimate preliminary effect sizes for DAPPER in reduction pain and depressive symptoms, 3) measure effect sizes and feasibility of measuring cytokines and heart rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Self-report pain >3 out of a 0 -10 scale that has lasted longer than 3 months and keeps subjects from doing at least one activity that subjects would like to do
* Self-Identify as African American/Black female
* Live in a community dwelling
* Score a 5 or higher on the PHQ-9 (depression measure) at least two times during a two week period (screening call and then at first data collection visit)
* Must be pre-frail (one or two criteria on frailty phenotype) or frail (three or more of the criteria on frailty phenotype)
* One ADL or IADL limitation

Exclusion Criteria:

* Hospitalized > 3 times in the last year
* Participating in physical therapy
* Have a terminal diagnosis (<1 year expected survival)
* > moderate intellectual impairment (5-7 errors) based on the Short Portable Mental Status Questionnaire (SPMSQ)
* Unable to speak or understand English

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janiece L Taylor, PhD, Principal Investigator — Johns Hopkins School of Nursing; Catherine Clair, MHS, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor JL, Clair CA, Lee JW, Atkins S, Riser TJ, Szanton SL, McCoy MC, Thorpe RJ Jr, Wang C, Gitlin LN. A protocol for a wait list control trial of an intervention to improve pain and depressive symptoms among middle-aged and older African American women. Contemp Clin Trials. 2023 Sep;132:107299. doi: 10.1016/j.cct.2023.107299. Epub 2023 Jul 20. PMID 37478967
- [Result] Taylor JL, Clair CA, Gitlin LN, Atkins S, Bandeen-Roche K, Abshire Saylor M, Hladek MD, Riser TJ, Thorpe RJ Jr, Szanton SL. Acceptability and Feasibility of a Pain and Depressive Symptoms Management Intervention in Middle-Aged and Older African American Women. Innov Aging. 2023 Sep 8;7(10):igad096. doi: 10.1093/geroni/igad096. eCollection 2023. PMID 38094930
- Available data/document: Study Protocol: 37478967 — https://pubmed.ncbi.nlm.nih.gov/37478967/
- Available data/document: Outcomes Manuscript: 38094930 — https://pubmed.ncbi.nlm.nih.gov/38094930/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Wait List Control Arm
Started | 17 | 17
Completed | 13 | 10
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Wait List Control Arm | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (11) | 64.6 (10.3) | 64.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity as Assessed by the Patient Reported Outcomes Measurement Information System (PROMIS)
Description: The PROMIS Intensity is used to measure pain intensity on a scale of 0-10. Higher scores indicate more pain intensity.
Time Frame: Baseline and 12 weeks
Population: A total of 23 participants completed the intervention. Participants who completed this measure at baseline (pre intervention) and post intervention (12 + weeks), (13 participants in the intervention group and 10 in the control group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 13 | 10
score on a scale
  Baseline | 6.75 (2.18) | 7.29 (1.57)
  12 weeks | 6.64 (1.80) | 7.00 (1.35)

2. Primary Outcome: Depressive Symptoms as Assessed by the Patient Health Questionnaire 9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9) includes 9 questions related to the Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnostic criteria for major depression. The PHQ-9 scores range from 0-27. Higher scores indicate more depressive symptoms.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 13 | 10
score on a scale
  Baseline | 12.25 (3.13) | 11.53 (4.78)
  12 weeks | 8.36 (4.43) | 11.43 (4.67)

3. Secondary Outcome: Interleukin (IL)-6 in Saliva (pg/ml)
Description: An decrease in IL 6 indicates a decrease in this inflammatory marker.
Time Frame: Baseline and 12 weeks
Population: Due to the COVID 19 pandemic, not all saliva samples were collected and not all samples had sufficient saliva.
Measure: Mean (Standard Deviation); unit: picograms/millilitre
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 10 | 4
picograms/millilitre
  Baseline | 7.97 (6.22) | 8.19 (3.66)
  12 weeks | 5.12 (5.31) | 7.54 (3.88)

4. Secondary Outcome: Interleukin (IL)-8 in Saliva (pg/ml)
Description: A decrease indicates a decrease IL8 , which is an inflammatory marker.
Time Frame: Pre intervention , Post intervention 12 weeks for Intervention arm
Population: Due to the COVID 19 pandemic, not all saliva samples were collected and not all samples had sufficient saliva.
Measure: Mean (Standard Deviation); unit: picograms/millilitre
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 10 | 4
picograms/millilitre
  Pre intervention | 1780.22 (1629.85) | 2847.77 (1583.21)
  Post intervention 12 weeks | 1305.79 (1618.97) | 1805.99 (1613.66)

5. Secondary Outcome: Interleukin (IL)-1 Beta in Saliva (pg/ml)
Description: A change in IL-1beta indicates a change in this cytokine or protein.
Time Frame: Baseline and Post intervention 12 weeks for intervention arm. Baseline for wait list control.
Population: Due to the COVID 19 pandemic, not all saliva samples were collected and not all samples had sufficient saliva.
Measure: Mean (Standard Deviation); unit: picograms/millilitre
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 10 | 4
picograms/millilitre
  Pre intervention | 154.7 (90.37) | 564.35 (571.66)
  Post intervention 12 weeks | 247.47 (379.06) | 347.73 (357.62)

6. Secondary Outcome: Tumor Necrosis Factor (TNF)-Alpha in Saliva (pg/ml)
Description: Tumor necrosis factor (TNF)-alpha in saliva (pg/ml). TNF-alpha is a cytokine that signals inflammation in the body. Higher levels indicate there may be more inflammation.
Time Frame: Baseline and post intervention (12 weeks ) for intervention arm. Baseline only (wait list control arm)
Population: Due to the COVID 19 pandemic not all saliva samples were collected and there was insufficient amount of saliva for some of the samples.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 10 | 4
pg/ml
  Pre intervention | 5.09 (7.57) | 7.66 (4.32)
  Post intervention 12 weeks | 3.56 (3.84) | 4.68 (2.94)

7. Other Pre Specified Outcome: Physical Function as Assessed by the Katz Activities of Daily Living (ADL)
Description: The Katz Activities of daily living (ADL) is used measure physical function through ability to perform activities of daily living. Score ranges are from 0-6 with 6 indicating full function and a score of 2 or less indicating severe functional impairment.
Time Frame: Baseline
Population: This was part of the inclusion criteria.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 17 | 17
score on a scale | 2.7 (1.8) | 2.6 (1.7)

8. Other Pre Specified Outcome: Physical Function as Assessed by the Lawton's Instrumental Activities of Daily Living (IADL)
Description: Lawton's Instrumental Activities of Daily Living (IADL) measures instrumental activities of daily living as a measure of physical function. The scores range from 0-8 with higher scores indicating better physical function.
Time Frame: Baseline
Population: This was measured as part of screening criteria to participate in the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 17 | 17
score on a scale | 3.2 (1.8) | 3.1 (1.7)

9. Other Pre Specified Outcome: Frailty as Assessed by the Frail Scale
Description: The Frail Scale is used to measure frailty. The scores range from 0-17 with higher scores indicating more frailty.
Time Frame: Baseline
Population: We used this outcome as inclusion criteria versus a measured outcome pre and post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 17 | 17
score on a scale | 2.9 (0.7) | 2.8 (0.6)

10. Other Pre Specified Outcome: Change in Depressive Symptoms as Assessed by the PROMIS 57
Description: The Patient Reported Outcomes Measurement System (PROMIS)57 the Patient Reported Outcomes Measurement Information System (PROMIS) 57, which is includes an 8-item instrument that can be used to measure self-reported negative mood, view of self, and somatic symptoms. The score range for PROMIS 57 is 8-40. Higher scores indicate more depressive symptoms.
Time Frame: Nurse Visit 1 and Nurse Visit 8
Population: Data not collected. Investigators used the PhQ9 as the measure of depression for this study as opposed to PROMIS 57.
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Stress as Assessed by the Perceived Stress Scale (Intervention Group)
Description: The Perceived Stress Scale assesses a person's perceived stress levels. The scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Pre intervention, Post intervention 12 weeks
Population: Participants with data collected in the intervention group only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 10 | 0
score on a scale
  Pre intervention | 25 (8.0) |
  Post intervention 12 weeks | 22.2 (9.2) |

12. Other Pre Specified Outcome: Comorbid Conditions as Assessed by the Charlson Comorbidity Index
Description: The Charlson Comorbidity Index consists of 17 categories of chronic conditions and two subcategories for diabetes and liver disease. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. Up to 12 comorbidities with various weightings can result in a maximum score of 24. Score range 0-24.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 17 | 17
score on a scale | 3.8 (1.9) | 3.9 (2.0)

13. Other Pre Specified Outcome: Change in Social Engagement as Assessed by the Social Network Scale
Description: The Lubben Social Network Scale -6 is used to measure social engagement including family and friends. The scores range from 0 to 60 with higher scores indicating more social engagement.
Time Frame: Baseline, 12 weeks and 24 weeks
Population: This data has not been analyzed and was a potential outcome that we proposed in our protocol.
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Change in Self Efficacy as Assessed by the Coping and Self-Efficacy Scale
Description: The Coping and Self-Efficacy Scale is a 26 item scale used to measure coping and self efficacy. The scores on this instrument range from 0-260 with higher scores indicating more self efficacy.
Time Frame: Baseline and 12 weeks
Population: Participants with data collected in the intervention group only
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Change in Frailty as Assessed by the Frailty Phenotype Measure
Description: The Frailty Phenotype measure is used to determine if a person is robust (score of 0), pre-frail (score of 1 or 2), or frail (score of 3-5). total score range of 0-5.
Time Frame: Baseline and 12 weeks
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait List Control Arm
Number analyzed (Participants) | 13 | 13
score on a scale | 3.15 (0.55) | 3.29 (0.49)

ADVERSE EVENTS:
Time Frame: Up to 45 months
Arm/Group | Intervention Arm | Wait List Control Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04091347/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT04091347/ICF_001.pdf